CLINICAL TRIAL: NCT03270124
Title: A pragmatiC sTrategy to Promote actIVity and Enhance Quality of Life AFTER Transcatheter Aortic Valve Replacement (ACTIVE AFTER TAVR): A Pilot Study
Brief Title: A pragmatiC sTrategy to Promote actIVity and Enhance Quality of Life AFTER Transcatheter Aortic Valve Replacement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: Edwards Lifesciences (Industry)
Responsible Party: Principal Investigator, Brian Lindman, Associate Professor, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACTIVE AFTER TAVR
Record Dates: First submitted 2017-08-29; First posted 2017-09-01 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Aortic Valve Stenosis
Keywords: Aortic Valve Stenosis; Fitbit; iPAD; Physical Exercises; Quality of Life
MeSH Terms: conditions — Aortic Valve Stenosis; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No Resistance Exercise and No Activity Goal Arm (Active Comparator): Blinded use of Fitbit with no daily activity goal and no resistance exercises
  Interventions: Behavioral: Daily Activity Recording
- Resistance Exercise and Activity Goal Arm (Experimental): Unblinded use of Fitbit with a daily activity goal (steps per day) and resistance exercises
  Interventions: Behavioral: Daily Activity Goal; Behavioral: Resistance Exercises; Behavioral: Daily Activity Recording

INTERVENTIONS:
Behavioral: Daily Activity Goal — Patients are given a tailored daily activity goal in terms of steps per day for which to aim.
  Other Names: Resistance Exercise and Activity Goal Arm
  Arms: Resistance Exercise and Activity Goal Arm
Behavioral: Resistance Exercises — Patients will instructed to perform 3 different resistance exercises targeting muscles pertinent to activities of daily living on 6 out of 7 days a week.
  Other Names: Resistance Exercise and Activity Goal Arm
  Arms: Resistance Exercise and Activity Goal Arm
Behavioral: Daily Activity Recording — A Fitbit will be worn by all participants to record daily activity.

SUMMARY:
This study is being performed in patients who have undergone transcatheter aortic valve replacement (TAVR) for aortic stenosis. The goal is to obtain pilot and feasibility data on a novel post-procedure rehabilitation strategy, including a daily activity goal using a fitness tracking device (Fitbit Alta HR) and in-home resistance training exercises targeting muscles related to activities of daily living. We will evaluate the effect of these interventions on physical performance and several quality of life domains.

DETAILED DESCRIPTION:
The study will be conducted in three phases. Subjects who have been treated commercially with TAVR with a SAPIEN 3 valve and are being discharged to home will be eligible for Phase 1. Once consented prior to discharge, patients will complete the KCCQ, PROMIS Questionnaires, 5m walk, chair stand, and handgrip tests. During phase 1, all subjects will have a Fitbit and answer quality of life questions on the iPad about their activities and quality of life. After 30 days, the subject will return to complete the PROMIS Questionnaires, 5m walk, chair stand, balance tests, and handgrip tests, as well as a KCCQ. If the subject has consistently provided data throughout Phase 1, they will be asked to continue on to Phases 2 and 3 and complete a 6 minute walk test at this baseline visit. For Phase 2, subjects will be randomized to one of two arms. In one arm, they will have a daily activity goal and resistance exercises; in the other arm, there will not be a daily activity goal and no resistance exercises given. After 6 weeks, the subject will return to complete the 5m walk, 6 minute walk test, chair stand, balance tests, and handgrip tests, PROMIS Questionnaires, as well as a KCCQ. Five months after enrollment into Phase 2, subjects will be given a Fitbit to track their daily activity for 1 week (Phase 3). They will also complete a KCCQ, PROMIS Questionnaires, and end of study questionnaire.

ELIGIBILITY:
Inclusion Criteria:

Phase 1 - Starts after the TAVR procedure and prior to discharge • Patients treated commercially with TAVR with a SAPIEN 3 valve

Phases 2 and 3 - Starts at 30 day post-TAVR follow-up visit

• Patients enrolled in Phase 1

Exclusion Criteria:

Phase 1 - Starts after the TAVR procedure and prior to discharge

* Stroke during or immediately after the TAVR procedure prior to discharge
* Inability to walk
* Non-English speaking (because the mobile app and CAT questionnaires are only in English)
* Physical or neuropsychiatric limitations that would prevent proficient use of the study tools and successful completion of the physical and quality of life assessments. These limitations may include, but are not limited to: blindness, neuropathy, severe tremor or disabling motor deficit, cognitive impairment (documentation of dementia in the medical record), or illiteracy.
* Unwillingness or inability of the subject to provide informed consent for Phase 1 (no LARs allowed)
* Planned discharge from hospital to skilled nursing or rehabilitation facility

Phases 2 and 3 - Starts at 30 day post-TAVR follow-up visit

* All exclusion criteria from Phase 1 apply
* Stroke during Phase 1
* Residing in a skilled nursing facility at the 30 day post-TAVR follow-up visit
* Patients with unreliable use of the iPad mobile app or Fitbit during Phase 1 (e.g. not wearing the Fitbit at least 10 waking hours a day for at least 5 days a week)
* Unwillingness or inability of the subject to provide informed consent for Phases 2/3 (no LARs allowed)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2017-11-07 (Actual); Primary Completion 2020-03-24 (Actual); Study Completion 2020-03-25 (Actual)

PRIMARY OUTCOMES:
Average Daily Steps | Randomization to 6 weeks
  Average daily steps over the intervention period
Short Physical Performance Battery score | 6 week value, adjusted for baseline value
  Combination of gait speed, balance test, and chair-to-stand test at the end of the intervention
Quality of Life as measured with the KCCQ Overall Summary Score | 6 week value, adjusted for baseline value
  KCCQ overall summary score

SECONDARY OUTCOMES:
5 meter gait time at the end of the intervention period | Randomization to 6 weeks
  5 meter gait time at the end of the intervention period, adjusted for baseline
Chair Sit to Stand Test | 6 week value, adjusted for baseline value
  Time to complete 5 chair stands
Balance Test Score at the end of the intervention period | Randomization to 6 weeks
  Balance Test Score at the end of the intervention period, adjusted for baseline
6 minute walk | 6 week value, adjusted for baseline value
  6 minute walk distance at the end of the intervention period
Handgrip | 6 week value, adjusted for baseline value
  Handgrip strength
Average number of hours per day with 250 or more steps | Randomization to 6 weeks
  Average number of hours per day with 250 or more steps over the intervention period
Average Global Physical Health as assessed by the PROMIS Global Health 10 Short Form | Randomization to 6 weeks
  Average Global Physical Health as assessed by the PROMIS Global Health 10 Short Form over the intervention period
Average Global Mental Health as assessed by the PROMIS Global Health 10 Short Form | Randomization to 6 weeks
  Average Global Mental Health as assessed by the PROMIS Global Health 10 Short Form over the intervention period
Physical Function as assessed by the NIH PROMIS computerized adaptive test | Randomization to 6 weeks
  Physical Function as assessed by the NIH PROMIS computerized adaptive test, adjusted for baseline
Depression as assessed by the NIH PROMIS computerized adaptive test | Randomization to 6 weeks
  Depression as assessed by the NIH PROMIS computerized adaptive test, adjusted for baseline
Fatigue as assessed by the NIH PROMIS computerized adaptive test | Randomization to 6 weeks
  Fatigue as assessed by the NIH PROMIS computerized adaptive test, adjusted for baseline
Dyspnea as assessed by the NIH PROMIS computerized adaptive test | Randomization to 6 weeks
  Dyspnea as assessed by the NIH PROMIS computerized adaptive test, adjusted for baseline
Daily Active Minutes (total) | Randomization to 6 weeks
  Average daily active minutes (total)
Daily Active Minutes of Moderate to High Intensity | Randomization to 6 weeks
  Average daily minutes of moderate to high intensity
Sedentary Minutes | Randomization to 6 weeks
  Average daily sedentary minutes
Daily Steps | 6 weeks post baseline to end of study
  Average daily steps
Daily Active Minutes (total) | 6 weeks post baseline to end of study
  Average daily active minutes (total)
Daily Active Minutes of Moderate to High Intensity | 6 weeks post baseline to end of study
  Average daily active minutes of moderate to high intensity
Daily Sedentary Minutes | 6 weeks post baseline to end of study
  Average daily sedentary minutes
KCCQ Overall Summary Score | 6 weeks post baseline to end of study
  KCCQ overall summary score, adjusted for baseline
Global Physical Health | 6 weeks post baseline to end of study
  Global physical health as assessed by the PROMIS Global Health 10 Short Form, adjusted for baseline
Global Mental Health | 6 weeks post baseline to end of study
  Global mental health as assessed by the PROMIS Global Health 10 Short Form, adjusted for baseline

CONTACTS AND LOCATIONS:
Overall Officials: Brian R Lindman, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (5):
- United States (5):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Atlantic Health - Morristown Medical Center, Morristown, New Jersey
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lindman BR, Gillam LD, Coylewright M, Welt FGP, Elmariah S, Smith SA, McKeel DA, Jackson N, Mukerjee K, Cloud H, Hanna N, Purpura J, Ellis H, Martinez V, Selberg AM, Huang S, Harrell FE Jr. Effect of a pragmatic home-based mobile health exercise intervention after transcatheter aortic valve replacement: a randomized pilot trial. Eur Heart J Digit Health. 2021 Feb 4;2(1):90-103. doi: 10.1093/ehjdh/ztab007. eCollection 2021 Mar. PMID 34048509
- [Derived] Abraham LN, Sibilitz KL, Berg SK, Tang LH, Risom SS, Lindschou J, Taylor RS, Borregaard B, Zwisler AD. Exercise-based cardiac rehabilitation for adults after heart valve surgery. Cochrane Database Syst Rev. 2021 May 7;5(5):CD010876. doi: 10.1002/14651858.CD010876.pub3. PMID 33962483